CLINICAL TRIAL: NCT04364581
Title: Endometrial Preparation by Short Course of Letrozole Before Hysteroscopic Removal of Endocavitary Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS.19.06.685.R1.R2
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Myoma;Uterus
Keywords: Letrozole; Submucous myoma
MeSH Terms: conditions — Myofibroma | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole group (Active Comparator): Women will be treated with letrozole (5 mg daily) for 10 days before hysteroscopic intervention
  Interventions: Drug: Letrozole
- Placebo group (Placebo Comparator): Women will be treated with placebo for 10 days before hysteroscopic intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letrozole — Women will be treated with letrozole (5 mg daily) for 10 days before hysteroscopic intervention
  Other Names: Femara
  Arms: Letrozole group
Drug: Placebo — Women will be treated with placebo for 10 days before hysteroscopic intervention
  Arms: Placebo group

SUMMARY:
The aim of this study is to evaluate the effectiveness of short course of letrozole for endometrial preparation before hysteroscopic surgery for intracavitary lesions.

DETAILED DESCRIPTION:
In the cycle subsequent to hysteroscopic identification of an endouteine pathology, patients who fitted with the inclusion criteria will be randomly divided into two groups; letrozole group (study group) and placebo group (control group). The randomization will be a stratified randomization with permuted blocking (the block size is randomly permuted among 2, 4, and 6) within each stratum. The only stratification variable will be by type of endouterine pathology. The randomization will be balanced (using a 1:1 treatment ratio) and will be carried out by a nurse through sealed, unlabeled, opaque envelopes containing computer-generated random numbers. The study will be double-blind (the participants, caregivers and investigators will be blinded to block size and group assignment).

Women in the letrozole group will be treated with letrozole (5 mg daily) for 10 days before hysteroscopic intervention while women in the placebo group will be treated with placebo for 10 days before hysteroscopic intervention in the early follicular phase of a natural cycle. In both groups, monopolar hysteroscopic surgery with glycine (1.5%) as uterine distension media will be used. Precise records of the duration of each surgical procedure, from the insertion to the removal of the resectoscope will be done.

Measurements of inflow, outflow, and amount of distension liquid absorbed by the patient will be taken meticulously. Intraoperative bleeding will be defined as "light" when bleeding does not interfere with surgery, "moderate" when bleeding required the coagulation of vessels, and "severe" when hemorrhage required immediate suspension of hysteroscopy. At the end of surgery, surgeon satisfaction with endometrial preparation using Visual Analogue Scale (VAS) and quality of visualization of the uterine cavity will be compared. Postoperative complications will be defined as the appearance of any complications occurring from the termination of the surgery to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endouterine pathologies, identified by office diagnostic hysteroscopy during the early endometrial proliferative phase (cycle days 7 to 8)

Exclusion Criteria:

* Presence of large submucous (type I, type II) or endocavitary (type 0) fibroids (according to the European Society of Hysteroscopy Classification of Submucous Fibroids) with a diameter exceeding 4 cm, for which preoperative treatment with GnRH agonists is indicated.
* Hormonal therapies in the previous 8 weeks (including the drug of the study).
* Uterine and/or concomitant adnexal pathologies (including malignancy) for which hysteroscopic surgery was not considered either safe or the method to resolve the problem.
* Cardiovascular, hepatic, or renal impairment.
* Allergy to letrozole.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | Until 2 hours from the start of operation
  Time from start to end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yomna Ayman, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, MD, Study Director — Mansoura University; Rafik I Barakat, MD, Study Director — Mansoura University; Tarek A Shokir, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided